CLINICAL TRIAL: NCT00091975
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind, Multi-Center Study to Evaluate the Safety and Efficacy of Zemplar® Capsule in Reducing Serum Intact Parathyroid Hormone Levels in Chronic Kidney Disease Stage 5 Subjects on Hemodialysis or Peritoneal Dialysis
Brief Title: Zemplar® Capsule in Reducing Serum Intact Parathyroid Hormone Levels in Chronic Kidney Disease Stage 5 Subjects on Hemodialysis or Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M03-635
Record Dates: First submitted 2004-09-20; First posted 2004-09-22 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2006-07

CONDITIONS: Kidney Disease
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic | interventions — paricalcitol

INTERVENTIONS:
Drug: Zemplar Capsule

SUMMARY:
The objective of this study is to determine the safety and efficacy of Zemplar® Capsule versus placebo, in decreasing elevated intact parathyroid hormone levels in chronic kidney disease stage 5 subjects with secondary hyperparathyroidism on hemodialysis or peritoneal dialysis, while using the revised dose titration scheme.

ELIGIBILITY:
Inclusion Criteria

* Subject was at least 18 years of age, diagnosed with CKD Stage 5 and undergoing HD or PD.
* If female, subject was either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or was of childbearing potential and practicing 1 of the protocol specified methods of birth control, was not breastfeeding and had a negative serum pregnancy test prior to the Treatment Phase.
* For those subjects taking phosphate binders prior to the study, the subject had to have been on a stable (type and dose) phosphate binder at least 4 weeks prior to the Pretreatment Phase.
* For entry into the Pretreatment Phase, the subject must have had a calcium level <= 10.5 mg/dL and a CaxP level <= 65 mg2/dL2.
* For entry into the Treatment Phase, the subject must have had iPTH >= 300 pg/mL (determined by Nichols iPTH assay), a calcium level of 8.0 to 10.5 mg/dL, inclusive, and CaxP <= 65 mg2/dL2.
* Subject voluntarily signed and dated an informed consent, approved by an Institutional Review Board (IRB), after the nature of the study was explained and the subject had the opportunity to ask questions. The informed consent was signed before any study-specific procedures were performed or any medications were withheld.
* Additional criteria for HD subjects included the following: the subject was diagnosed with CKD Stage 5 and must have been on maintenance HD 3 times a week (TIW) for at least 2 months prior to the Screening Phase and was expected to remain on HD for the duration of the study.
* Additional criteria for PD subjects, included the following: the subject was diagnosed with CKD Stage 5 and must have been on continuous PD (either continuous cycling peritoneal dialysis [CCPD], continuous ambulatory peritoneal dialysis [CAPD], or a combination of the 2) 7 days per week for at least 2 months prior to the Screening Phase and was expected to remain on this PD regimen for the duration of the study.

Exclusion Criteria

* Subject had a history of an allergic reaction or significant sensitivity to drugs similar to the study drug.
* Subject received a partial parathyroidectomy within 1 year prior to the Screening Phase.
* Subject had acute renal failure within 3 months of the Screening Phase.
* Subject had chronic gastrointestinal disease, which in the investigator's opinion, may have resulted in clinically significant gastrointestinal malabsorption.
* Subject had taken aluminum-containing phosphate binders for > 3 weeks in the last 3 months prior to the Screening Phase, or required such medications for > 3 weeks in the study.
* Subject had a current malignancy (with the exception of basal or squamous cell carcinoma of the skin), or clinically significant liver disease, in the opinion of the investigator.
* Subject had a history of drug or alcohol abuse within 6 months prior to the Screening Phase.
* Subject had evidence of poor compliance with diet, medication or HD/PD that may have interfered, in the investigator's opinion, with adherence to the protocol.
* Subject had participated in any investigational drug or device study within 4 weeks prior to the Treatment Phase.
* Subject was taking calcitonin, maintenance IV or oral glucocorticoids, cinacalcet, bisphosphonates, vitamin D compounds (other than study drug), or other drugs that may have affected calcium or bone metabolism, other than females on stable estrogen and/or progestin therapy.
* Subject was known to be human immunodeficiency virus (HIV) positive.
* For any reason, subject was considered by the investigator to be an unsuitable candidate to receive Zemplar.
* Additional exclusion criteria for PD subjects, were: Subject had active peritonitis within 1 month prior to the Screening Phase; Subject had more than 1 episode of peritonitis within 4 months prior to the Screening Phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78
Dates: Start 2004-08

PRIMARY OUTCOMES:
The efficacy endpoint is achievement of two consecutive > or = 30% decreases from baseline in iPTH levels

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Williams, M.D., MPH, Study Director — Abbott
Locations (16):
- United States (16):
  - California Institute of Renal Research, San Diego, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Associates in Nephrology, Fort Meyers, Florida
  - University of Florida, Gainesville, Florida
  - Outcomes Research International, Inc., Hudson, Florida
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Washington University Medical Center, St Louis, Missouri
  - St. Louis University, St Louis, Missouri
  - Nea Research, Las Vegas, Nevada
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Northwestern Renal Clinic, INC., Portland, Oregon
  - Nephrology Associates, P.C., Nashville, Tennessee
  - Kidney Associates, PLLC, Houston, Texas
  - University of Texas Health Center at San Antonio, San Antonio, Texas

REFERENCES:
- See also: Product Information — http://www.humira.com/